CLINICAL TRIAL: NCT01369784
Title: Observational, Post-authorization, Cross-sectional Study to Evaluate the Prognostic Value of Clinical and Biological Factors in Patients With Refractory/Relapsed Diffuse Large B-cell Lymphoma
Brief Title: Prognostic Value of Clinical and Biological Factors in Patients With Refractory/Relapsed Diffuse Large B-cell Lymphoma
Acronym: PRO-R-IPI
Status: Completed | Type: Observational
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-R-IPI
Record Dates: First submitted 2011-02-23; First posted 2011-06-09 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B-cell Lymphoma; R-IPI
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- refractory/relapsed LDCBG: patients with refractory/relapsed diffuse large B-cell lymphoma

SUMMARY:
The purpose of this study is to evaluate the prognostic value of clinical and biological factors in patients with refractory/relapsed Diffuse Large B-Cell Lymphoma.

DETAILED DESCRIPTION:
The main aim of this study is to compare the prognostic value of R-IPI at diagnosis and relapse, relating it with the obtained response after second line

ELIGIBILITY:
* Age 18 > years old
* Patients with refractory/relapsed diffuse large B-cell lymphoma after first line treatment with rituximab, with or without transplantation. Patients must have finished a rescue treatment including rituximab
* Ability to understand and willingness to sign a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory/relapsed diffuse large B-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Panizo, PhD, Study Chair — Grupo Español de Linfomas/Trasplante Autólogo de Médula Ósea
Locations (56):
- Spain (56):
  - Hospital de Elda, Elda, Alicante
  - H. U. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall D'Hebrón, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - ICO-DYR, L'Hospitalet de Llobregat, Barcelona
  - Althaia, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - H. Sierrallana, Torrelavega, Cantabria
  - Hospital General del SAS de Jerez, Jerez de la Frontera, Cádiz
  - Institut Catalá d'Oncologia de Girona, Girona, Gerona
  - H.U. Virgen de las Nieves, Granada, Granada
  - Hospital Galdakao, San Sebastián, Guipuzcoa
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - C.H.U. A Coruña, A Coruña, La Coruña
  - H. Clínico U. Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital de León, León, León
  - Hospital Xeral, Lugo, Lugo
  - Hospital Universitario Arnau de Vilanova, Lleida, Lérida
  - H.U. Fundación Alcorcón, Alcorcón, Madrid
  - H.U.de Getafe, Getafe, Madrid
  - H. Severo Ochoa, Leganés, Madrid
  - H. Ramón y Cajal, Madrid, Madrid
  - H. U. La Princesa, Madrid, Madrid
  - H.G.U. Gregorio Marañón, Madrid, Madrid
  - H.U. La Paz, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - MD Anderson, Madrid, Madrid
  - Hospital Son Llatzer, Mallorca, Mallorca
  - H.U. Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Morales Messeguer, Murcia, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - H. Carlos Haya, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Complexo Hospitalario de Ourense, Ourense, Orense
  - Hospital Universitario Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - H. U. Central de Asturias, Oviedo, Principality of Asturias
  - H. Universitario de Salamanca, Salamanca, Salamanca
  - H. General de Segovia, Segovia, Segovia
  - H.U. Nuestra Señora de Valme, Seville, Sevilla
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - H. Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - H. Arnau de Vilanova, Valencia, Valencia
  - H. Clínico de Valencia, Valencia, Valencia
  - H. Dr. Peset, Valencia, Valencia
  - H. Río Hortega, Valladolid, Valladolid
  - Hospital Clínico Universitario Valladolid, Valladolid, Valladolid
  - H. Basurto, Bilbao, Vizcaya
  - H. Virgen de La Concha, Zamora, Zamora
  - H. Txagorritxu, Vitoria-Gasteiz, Álava
  - H. Nuestra Señora de Sonsoles, Ávila, Ávila

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out between April 2009 and January 2011 in Hematology Departments of 56 Spanish Hospitals
Groups:
- Refractory/Relapsed LDCBG (Diffuse Large-B-cell Lymphoma): patients with refractory/relapsed diffuse large B-cell lymphoma
Period: Overall Study
Arm/Group | Refractory/Relapsed LDCBG (Diffuse Large-B-cell Lymphoma)
Started | 158
Completed | 146
Not Completed | 12
Not completed — Protocol Violation | 12

BASELINE CHARACTERISTICS:
Population: 12 patients were not included in the data analysis for not fulfilling selection criteria
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 78
Ann Arbor Staging [Number; unit: participants] — Ann Arbor=I: Best condition Ann Arbor=IV: Worst condition
  participants
    I | 6
    II | 20
    III | 37
    IV | 83
ECOG Performance Status (Eastern Cooperative Oncology Group Performance Status) [Number; unit: participants] — ECOG=0: Fully active, able to carry on all pre-disease performance without restriction ECOG=5: Exitus
  participants
    ECOG 0 | 48
    ECOG 1 | 55
    ECOG 2 | 25
    ECOG 3 | 15
    ECOG 4 | 3

OUTCOME MEASURES:

1. Primary Outcome: R-IPI Index (Revised International Prognostic Index)
Description: Data will be recorded from diagnosis to second line response, an expected average of 7 months
Time Frame: At diagnoses
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Very good prognosis (0) | 3.4
  Good prognosis (1,2) | 32.2
  Poor prognosis (3,4,5) | 64.4

2. Secondary Outcome: Bcl-2 Expression
Description: immunohistochemical reaction of cells with Bcl-2 antibody
Time Frame: At diagnosis
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 54.1
  Negative | 8.9
  Not available | 37.0

3. Secondary Outcome: Bcl-2 Expression
Description: immunohistochemical reaction of cells with Bcl-2 antibody
Time Frame: At the beginning of the 2nd line of treatment
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
participants
  Positive | 30
  Negative | 5
  Not Available | 111

4. Secondary Outcome: Bcl-6 Expression
Description: immunohistochemical reaction of cells with Bcl-6 antibody
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
participants
  Positive | 63
  Negative | 20
  Not available | 63

5. Secondary Outcome: Bcl-6 Expression
Description: immunohistochemical reaction of cells with Bcl-6 antibody
Time Frame: At the beginning of the second line of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 14.4
  Negative | 7.5
  Not available | 78.1

6. Primary Outcome: R-IPI Index (Revised International Prognostic Index)
Description: The IPI is based on the evaluation of 5 clinical factors: age > 60 years Ann Arbor stage III or IV disease > 1 extra nodal site European Cooperative Oncology Group performance status (ECOG PS) _ 2, increased serum LDH (lactate dehydrogenase) levels Revised IPI (R-IPI) evaluates the same parameters, but groups them differently to form 3 prognostic groups of patients with significantly different progression-free survival and overall survival outcomes.
Time Frame: At the beginning of the 2nd line of treatment, an average of 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of patients
  Very good prognosis (0) | 9.6
  Good prognosis (1,2) | 47.3
  Poor prognosis (3,4,5) | 43.2

7. Secondary Outcome: p-53 Expression
Description: immunohistochemical reaction of cells with p-53 antibody
Time Frame: At diagnosis
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 12.3
  Negative | 10.3
  Not available | 77.4

8. Secondary Outcome: p53 Expression
Description: immunohistochemical reaction of cells with p-53 antibody
Time Frame: At the beginning of the 2nd line of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 5.5
  Negative | 4.8
  Not available | 89.7

9. Secondary Outcome: Multiple Myeloma Oncogene 1 (MUM-1) Expression
Description: immunohistochemical reaction of cells with MUM-1 antibody
Time Frame: At diagnosis
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 16.4
  Negative | 10.3
  Not available | 73.3

10. Secondary Outcome: MUM-1 Expression
Description: immunohistochemical reaction of cells with MUM-1 antibody
Time Frame: At the beginning of the 2nd line of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of participants
  Positive | 5.5
  Negative | 5.5
  Not available | 89.0

11. Secondary Outcome: Eastern Cooperative Oncology Group Performance Status (ECOG) Performance Status
Description: ECOG=0: Fully active, able to carry on all pre-disease performance without restriction ECOG=5: Exitus
Time Frame: At the beginning of the 2nd line of treatment
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
participants
  ECOG 0 | 56
  ECOG 1 | 54
  ECOG 2 | 22
  ECOG 3 | 12
  ECOG 4 | 2

12. Secondary Outcome: Ann Arbor Staging
Description: Ann Arbor=I: Best condition Ann Arbor=IV: Worst condition
Time Frame: At the beginning of the 2nd line of treatment
Measure: Number; unit: percentage of patients
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
percentage of patients
  I | 12.3
  II | 21.9
  III | 19.9
  IV | 45.9

13. Secondary Outcome: Response to First Line of Treatment
Description: Complete Response (CR), Disappearance of all target lesions for at least 8 weeks.
  Partial response (PR): At least a 50% dicrease in the sum of the products of two measurements (the maximum diameter of a tumor and the largest diameter perpendicular to this maximum diameter) of 6 biggest individual tumors. Not increased of measure of other tumors, spleen or liver Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive Disease (PD): At least a 50% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions during or at the end of the treatment.
Time Frame: After first line treatment
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 146
participants
  Complete response | 58
  Uncertain complete response | 5
  Partial response | 52
  Stable disease | 10
  Progressive disease | 21

14. Secondary Outcome: Response to Second Line of Treatment
Description: as for outcome 13
Time Frame: After second line of treatment
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Complete response | 46
  Uncertain complete response | 15
  Partial response | 27
  Stable disease | 9
  Progressive disease | 38
  Not evaluated | 10

15. Primary Outcome: Predictive Value of R-IPI at Diagnosis
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Global response to 2nd line + very good prognos | 4
  No global response to 2nd line + very good prognos | 1
  Global response to 2nd line + good prognosis | 28
  No global response to 2nd line + good prognosis | 19
  Global response to 2nd line + poor prognosis | 56
  No global response to 2nd line + poor prognosis | 37
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.812, Fisher Exact

16. Secondary Outcome: Relationship Between Global Response Rate to 2nd (Second) Line of Treatment and Bcl-2 Expression at Diagnosis
Description: Global response rate was assessed using the National Cancer Institute-sponsored Working Group guidelines. Responses are: complete response, partial response, stable disease, progression and relapse
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Global response to 2nd line + Bcl-2 + | 50
  Global response to 2nd line + Bcl-2 - | 8
  No global response to 2nd line + Bcl-2 + | 28
  No global response to 2nd line + Bcl-2 - | 5
  Global response to 2nd line +Bcl-2 ND | 30
  No global response to 2nd line + Bcl-2 ND | 24
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.612, Chi-squared

17. Secondary Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and Bcl-6 Expression at Diagnosis
Description: as for outcome 16
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Global response to 2nd line + Bcl-6 + | 34
  Global response to 2nd line + Bcl-6 - | 14
  Global response to 2nd line + Blc-6 ND | 40
  No global response to 2nd line + Bcl-6 + | 28
  No global response to 2nd line + Bcl-6 - | 6
  No global response to 2nd line + Bcl-6 ND | 23
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.402, Chi-squared

18. Secondary Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and p53 Expression at Diagnosis
Description: as for outcome 16
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Global response to 2nd line + p53+ | 13
  Global response to 2nd line + p53- | 8
  No global response to 2nd line + p53+ | 5
  No global response to 2nd line + p53- | 6
  Global response to 2nd line + p53 ND | 67
  Global response to 2nd line + p53 - ND | 46
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.557, Chi-squared

19. Secondary Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and Multiple Myeloma Oncogene 1 (MUM1) Expression at Diagnosis
Description: as for outcome 16
Time Frame: At diagnosis
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 145
participants
  Global response to 2nd line + MUM1 + | 17
  Global response to 2nd line + MUM1 - | 6
  No global response to 2nd line + MUM1 + | 7
  No global response to 2nd line + MUM1 - | 8
  Global response to 2nd line + MUM1 ND | 65
  No global response to 2nd line + MUM1 ND | 42
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.234, Chi-squared

20. Post Hoc Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and Absolute Lymphocyte Count on Relapse
Description: as for outcome 16
Time Frame: At relapse
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 142
participants
  Global response to 2nd line + lymphocyte <1 | 40
  Global response to 2nd line + lymphocyte >=1 | 47
  No global response to 2nd line + lymphocyte <1 | 35
  No global response to 2nd line + lymphocyte >=1 | 20
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.057, Fisher Exact

21. Post Hoc Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and Lymphocyte/Monocyte Rate on Relapse
Description: as for outcome 16
Time Frame: At relapse
Measure: Number; unit: participants
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 141
participants
  Global response to 2nd line + ratio <=2.6 | 46
  Global response to 2nd line + ratio >2.6 | 40
  No global response to 2nd line + ratio <=2.6 | 37
  No global response to 2nd line + ratio >2.6 | 18
Statistical Analysis 1: Comparison: Refractory/Relapsed LDCBG; Test type: Superiority or Other; p = 0.117, Fisher Exact

22. Post Hoc Outcome: Relationship Between Global Response Rate to 2nd Line of Treatment and Beta-2 Microglobulin at Relapse
Description: as for outcome 16
Time Frame: At relapse
Measure: Mean (Standard Deviation); unit: mg/100ml
Arm/Group | Refractory/Relapsed LDCBG
Number analyzed (Participants) | 88
mg/100ml
  Global response to 2nd line | 2.47 (1.51)
  No global response to 2nd line | 2.41 (1.51)

ADVERSE EVENTS:
Arm/Group | Refractory/Relapsed LDCBG
Serious Adverse Events (participants affected / at risk) | 18/146
Other Adverse Events (participants affected / at risk) | 44/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refractory/Relapsed LDCBG (N=146)
Neutropenia (Blood and lymphatic system disorders) | 7
Leucopenia (Blood and lymphatic system disorders) | 6
Trombocitopenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Refractory/Relapsed LDCBG (N=146)
Fatigue (General disorders) | 17
Gastrointestinal symptoms (Gastrointestinal disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No